CLINICAL TRIAL: NCT01814748
Title: A Phase III, Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate the Safety and Efficacy of MK-3102 in ≥18 and <45 Year-Old Subjects With Type 2 Diabetes Mellitus and Inadequate Glycemic Control
Brief Title: A Study of the Safety and Efficacy of Omarigliptin (MK-3102) in ≥18 and <45 Year-Old Participants With Type 2 Diabetes Mellitus and Inadequate Glycemic Control (MK-3102-028)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3102-028; 2012-004303-12 (EudraCT Number)
Record Dates: First submitted 2013-03-18; First posted 2013-03-20 (Estimated); Results first posted 2016-07-18 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-08

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus; Diabetes Mellitus, Type 2; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases; Metformin; Hypoglycemic Agents; Pharmacologic Actions; Therapeutic Uses
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases | interventions — 2-(2,5-difluorophenyl)-5-(2-(methylsulfonyl)-2,6-dihydropyrrolo(3,4-c)pyrazol-5(4H)-yl)tetrahydro-2H-pyran-3-amine; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Omarigliptin 25 mg (Experimental): Omarigliptin 25 mg, once weekly, for 24 weeks. Open-label metformin daily was to be initiated for participants meeting protocol-specified glycemic criteria, but was otherwise prohibited.
  Interventions: Drug: Omarigliptin; Drug: Metformin
- Placebo (Placebo Comparator): Placebo to omarigliptin, once weekly, for 24 weeks. Open-label metformin daily was to be initiated for participants meeting protocol-specified glycemic criteria, but was otherwise prohibited.
  Interventions: Drug: Placebo to omarigliptin; Drug: Metformin

INTERVENTIONS:
Drug: Omarigliptin — Omarigliptin 25 mg capsule administered orally once weekly
  Other Names: MK-3102
  Arms: Omarigliptin 25 mg
Drug: Placebo to omarigliptin — Matching placebo to omarigliptin 25 mg capsule administered orally once weekly
  Arms: Placebo
Drug: Metformin — Open-label metformin (dosed daily according to the country-specific product label) was to be initiated for participants meeting protocol-specified glycemic criteria, but was otherwise prohibited.
  Other Names: Fortamet®; Glucophage®; Glucophage® XR; Glumetza®; Riomet®; Metgluco®; Glycoran®

SUMMARY:
This study will examine the safety and efficacy of once-weekly omarigliptin in participants 18 to <45 years of age with Type 2 diabetes mellitus and inadequate glycemic control. The study hypothesis is that treatment with omarigliptin compared with placebo provides greater reduction in hemoglobin A1c (A1C) in participants after 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Has type 2 diabetes mellitus
* Currently not on an antihyperglycemic agent (AHA) for at least the past 12 weeks and has not been treated with omarigliptin at any time prior to study participation
* Participant is one of the following:

  1. Male
  2. Female who is not of reproductive potential
  3. Female of reproductive potential who agrees to remain abstinent from heterosexual activity or use (or have her partner use) 2 acceptable methods of contraception to prevent pregnancy during the study and for 21 days after the last dose of study drug

Exclusion Criteria:

* History of type 1 diabetes mellitus or a history of ketoacidosis
* History of hypersensitivity to dipeptidyl-peptidase-4 (DPP-4) inhibitor
* Currently participating in or has participated in a clinical trial in the past 12 weeks
* Is on a weight loss program and not in the maintenance phase; has been on a weight loss medication in the past 6 months; or has undergone bariatric surgery within 12 months prior to study participation
* Has undergone a surgical procedure within 4 weeks of study participation or has planned major surgery during the study
* Is on or likely to require treatment for ≥14 consecutive days or repeated courses of pharmacologic doses of corticosteroids
* Is currently being treated for hyperthyroidism or is on thyroid replacement therapy and has not been on a stable dose for at least 6 weeks
* Is expecting to undergo hormonal therapy in preparation to donate eggs during the study, including 21 days following the last dose of study drug
* History of active liver disease (other than non-alcoholic hepatic steatosis) including chronic active hepatitis B or C, primary biliary cirrhosis, or symptomatic gallbladder disease
* Has human immunodeficiency virus (HIV)
* Has had new or worsening coronary heart disease or congestive heart failure within the past 3 months, or has any of the following disorders within the past 3 months:

  1. Acute coronary syndrome
  2. Coronary artery intervention
  3. Stroke or transient ischemic neurological disorder
* Has poorly controlled hypertension
* History of malignancy ≤5 years prior to study participation, except for basal cell or squamous cell skin cancer or in situ cervical cancer
* Has a hematological disorder (such as aplastic anemia, myeloproliferative or myelodysplastic syndromes, thrombocytopenia)
* Has a positive urine pregnancy test
* Pregnant or breastfeeding, or is expecting to conceive during the study, including 21 days following the last dose of study drug
* User of recreational or illicit drugs or has had a recent history of drug abuse. Routinely consumes >2 alcoholic drinks per day or >14 alcoholic drinks per week, or engages in binge drinking.
* Has donated blood products or has had a phlebotomy (>300 mL) within 8 weeks of study participation, or intends to donate blood products during the study or has received, or is anticipated to receive, blood products within 12 weeks of study participation or during the study
* Has a clinically significant electrocardiogram abnormality

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 203 (Actual)
Dates: Start 2013-05-03 (Actual); Primary Completion 2015-09-14 (Actual); Study Completion 2015-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Gantz I, Sokolova L, Jain L, Iredale C, O'Neill EA, Wei Z, Lam R, Suryawanshi S, Kaufman KD, Engel SS, Lai E. Use of Prohibited Medication, a Potentially Overlooked Confounder in Clinical Trials: Omarigliptin (Once-weekly DPP-4 Inhibitor) Monotherapy Trial in 18- to 45-year-olds. Clin Ther. 2017 Oct;39(10):2024-2037. doi: 10.1016/j.clinthera.2017.08.009. Epub 2017 Sep 18. PMID 28923291

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Omarigliptin 25 mg | Placebo
Started | 102 | 101
Completed | 94 | 94
Not Completed | 8 | 7
Not completed — Lost to Follow-up | 1 | 2
Not completed — Study site terminated by sponsor | 1 | 1
Not completed — Withdrawal by Subject | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Omarigliptin 25 mg | Placebo | Total
Number analyzed (Participants) | 102 | 101 | 203
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.8 (4.7) | 39.5 (4.5) | 39.2 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 41 | 76
  Male | 67 | 60 | 127
Hemoglobin A1c (A1C) [Mean (Standard Deviation); unit: Percent] | 7.9 (0.8) | 8.1 (0.9) | 8.0 (0.8)
2-hour post-meal glucose (2-hr PMG) [Mean (Standard Deviation); unit: mg/dL] — Participants with available data at baseline: Omarigliptin, n=98; Placebo, n=101; Total, n=199
  mg/dL | 204.9 (55.1) | 217.3 (67.7) | 211.2 (62.0)
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mg/dL] | 164.0 (38.9) | 167.8 (40.6) | 165.9 (39.7)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in A1C at Week 24
Description: A1C (%) is used to report average blood glucose levels over prolonged periods of time.
  The unexpected absence of a treatment effect in this study led to investigations that included measurement of metformin levels in available samples collected for future research during the study. Of the 92 participants with samples who had not been rescued with metformin, 57% (25/44) in the placebo group and 29% (14/48) in the omarigliptin group had detectable metformin, indicating the use of metformin that was prohibited by the protocol. The use of metformin prohibited by the protocol was without investigator knowledge and is a confounding factor impacting the ability to draw any conclusions regarding the efficacy results from this study.
Time Frame: Baseline and Week 24
Population: Full analysis set (FAS) population comprised all participants who received at least one dose of study treatment and had a baseline measurement or a post-randomization measurement for the analysis endpoint.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Omarigliptin 25 mg | Placebo
Number analyzed (Participants) | 102 | 101
Percent | -0.33 [-0.60 to -0.06] | -0.45 [-0.72 to -0.18]
Statistical Analysis 1: Comparison: Omarigliptin 25 mg vs Placebo; Test type: Superiority or Other; p = 0.535, Constrained longitudinal data analysis; Terms for treatment, time, and the interaction of time by treatment, with the constraint that the mean baseline is the same for all treatment groups; Difference in least squares means = 0.12, 95% CI 2-sided [-0.26 to 0.49]

2. Primary Outcome: Percentage of Participants Who Experienced at Least One Adverse Event (AE)
Description: An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study. Data presented exclude data following the initiation of glycemic rescue.
  The safety database was analyzed in a standard fashion in the all participants as treated (APaT) population for all participants who took at least one dose of study medication. This analysis may have been confounded by the use of metformin prohibited by the protocol (see efficacy results description above).
Time Frame: Up to Week 27
Population: APaT population included all randomized participants who received at least one dose of study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Omarigliptin 25 mg | Placebo
Number analyzed (Participants) | 102 | 101
Percentage of participants | 39.2 | 39.6
Statistical Analysis 1: Comparison: Omarigliptin 25 mg vs Placebo; Test type: Superiority or Other; Difference in percent = -0.4, 95% CI 2-sided [-13.8 to 13.0]

3. Primary Outcome: Percentage of Participants Who Discontinued Study Drug Due to an AE
Description: An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study. Data presented exclude data following the initiation of glycemic rescue.
  The safety database was analyzed in a standard fashion in the APaT population for all participants who took at least one dose of study medication. This analysis may have been confounded by the use of metformin prohibited by the protocol (see efficacy results description above).
Time Frame: Up to Week 24
Population: APaT population included all randomized participants who received at least one dose of study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Omarigliptin 25 mg | Placebo
Number analyzed (Participants) | 102 | 101
Percentage of participants | 0.0 | 2.0
Statistical Analysis 1: Comparison: Omarigliptin 25 mg vs Placebo; Test type: Superiority or Other; Difference in percent = -2.0

4. Secondary Outcome: Change From Baseline in 2-hr PMG at Week 24
Description: Blood glucose was measured 120 minutes from start of meal.
  The unexpected absence of a treatment effect in this study led to investigations that included measurement of metformin levels in available samples collected for future research during the study. Of the 92 participants with samples who had not been rescued with metformin, 57% (25/44) in the placebo group and 29% (14/48) in the omarigliptin group had detectable metformin, indicating the use of metformin that was prohibited by the protocol. The use of metformin prohibited by the protocol was without investigator knowledge and is a confounding factor impacting the ability to draw any conclusions regarding the efficacy results from this study.
Time Frame: Baseline and Week 24
Population: FAS population comprised all participants who received at least one dose of study treatment and had a baseline measurement or a post-randomization measurement for the analysis endpoint.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Omarigliptin 25 mg | Placebo
Number analyzed (Participants) | 100 | 101
mg/dL | -11.3 [-26.1 to 3.5] | -15.5 [-30.6 to -0.3]
Statistical Analysis 1: Comparison: Omarigliptin 25 mg vs Placebo; Test type: Superiority or Other; p = 0.685, Constrained longitudinal data analysis; [statistical method as in outcome 1, analysis 1]; Difference in least squares means = 4.2, 95% CI 2-sided [-16.1 to 24.4]

5. Secondary Outcome: Change in Baseline in FPG at Week 24
Description: Blood glucose was measured on a fasting basis.
  The unexpected absence of a treatment effect in this study led to investigations that included measurement of metformin levels in available samples collected for future research during the study. Of the 92 participants with samples who had not been rescued with metformin, 57% (25/44) in the placebo group and 29% (14/48) in the omarigliptin group had detectable metformin, indicating the use of metformin that was prohibited by the protocol. The use of metformin prohibited by the protocol was without investigator knowledge and is a confounding factor impacting the ability to draw any conclusions regarding the efficacy results from this study.
Time Frame: Baseline and Week 24
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Omarigliptin 25 mg | Placebo
Number analyzed (Participants) | 102 | 101
mg/dL | -5.0 [-14.6 to 4.6] | -1.3 [-11.2 to 8.5]
Statistical Analysis 1: Comparison: Omarigliptin 25 mg vs Placebo; Test type: Superiority or Other; p = 0.586, Constrained longitudinal data analysis; [statistical method as in outcome 1, analysis 1]; Difference in least squares means = -3.7, 95% CI 2-sided [-17.1 to 9.7]

6. Secondary Outcome: Percentage of Participants Attaining A1C Glycemic Goals of <7.0% at Week 24
Description: Percentage of participants was estimated using standard multiple imputation techniques (constrained longitudinal data analysis [cLDA] model). Within-group confidence intervals (CIs) were calculated via the Wilson score method.
  The unexpected absence of a treatment effect in this study led to investigations that included measurement of metformin levels in available samples collected for future research during the study. Of the 92 participants with samples who had not been rescued with metformin, 57% (25/44) in the placebo group and 29% (14/48) in the omarigliptin group had detectable metformin, indicating the use of metformin that was prohibited by the protocol. The use of metformin prohibited by the protocol was without investigator knowledge and is a confounding factor impacting the ability to draw any conclusions regarding the efficacy results from this study.
Time Frame: Week 24
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Omarigliptin 25 mg | Placebo
Number analyzed (Participants) | 102 | 101
Percentage of participants | 33.5 [24.7 to 43.7] | 34.0 [25.1 to 44.1]
Statistical Analysis 1: Comparison: Omarigliptin 25 mg vs Placebo; Test type: Superiority or Other; Mietinnen and Nurminen; Between-group rate difference = -0.4, 95% CI 2-sided [-14.0 to 13.1]

7. Secondary Outcome: Percentage of Participants Attaining A1C Glycemic Goals of <6.5% (48 mmol/Mol) at Week 24
Description: Percentage of participants was estimated using standard multiple imputation techniques (cLDA). Within-group CIs were calculated via the Wilson score method.
  The unexpected absence of a treatment effect in this study led to investigations that included measurement of metformin levels in available samples collected for future research during the study. Of the 92 participants with samples who had not been rescued with metformin, 57% (25/44) in the placebo group and 29% (14/48) in the omarigliptin group had detectable metformin, indicating the use of metformin that was prohibited by the protocol. The use of metformin prohibited by the protocol was without investigator knowledge and is a confounding factor impacting the ability to draw any conclusions regarding the efficacy results from this study.
Time Frame: Week 24
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Omarigliptin 25 mg | Placebo
Number analyzed (Participants) | 102 | 101
Percentage of participants | 21.7 [14.5 to 31.1] | 17.6 [11.3 to 26.5]
Statistical Analysis 1: Comparison: Omarigliptin 25 mg vs Placebo; Test type: Superiority or Other; Mietinnen and Nurminen; Between-group rate difference = 4.0, 95% CI 2-sided [-7.4 to 15.5]

8. Secondary Outcome: Percentage of Participants Who Required Glycemic Rescue by Week 24
Description: Participants exceeding pre-specified glycemic thresholds after starting the double-blind treatment period may have received rescue therapy (per protocol) with open-label metformin initiated by the investigator.
  This analysis may have been confounded by the use of metformin prohibited by the protocol (see efficacy results description above).
Time Frame: Up to Week 24
Population: All randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Omarigliptin 25 mg | Placebo
Number analyzed (Participants) | 102 | 101
Percentage of participants | 10.8 | 12.9

ADVERSE EVENTS:
Time Frame: Up to 27 weeks; Serious adverse events (SAEs) were collected up to 24 weeks during treatment + 3 week follow-up, non-serious adverse events (NSAEs) were collected up to 24 weeks during treatment
Description: SAEs include data after glycemic rescue; NSAEs exclude data after glycemic rescue. Investigations performed by the Sponsor revealed that many participants had used a prohibited antihyperglycemic agent-metformin (i.e., not as rescue medication; see efficacy results description above).
Arm/Group | Omarigliptin 25 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 1/102 | 3/101
Other Adverse Events (participants affected / at risk) | 10/102 | 7/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omarigliptin 25 mg (N=102) | Placebo (N=101)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omarigliptin 25 mg (N=102) | Placebo (N=101)
Nausea (Gastrointestinal disorders) | 6 (6) | 2 (2)
Headache (Nervous system disorders) | 6 (6) | 6 (6)

LIMITATIONS AND CAVEATS:
Investigations indicate that the presence of metformin in future biomedical research (FBR) samples from non-rescued participants was due to participant self-administration of metformin outside of the protocol and without investigator knowledge.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.